CLINICAL TRIAL: NCT04017013
Title: Therapeutic Efficacy of Intravenous Lidocaine Infusion Compared With Epidural Analgesia for Postoperative Pain Control in Adult Patients Undergoing Major Abdominal Surgery: Non-Inferiority Clinical Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Collaborators: IPS Universitaria-Universidad de Antioquia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIIU 2001-15550
Record Dates: First submitted 2019-06-19; First posted 2019-07-12 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-05

CONDITIONS: Pain, Postoperative; Opioid Use
Keywords: Pain; Abdominal Surgery; Epidural analgesia; lidocaine
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Analgesia, Epidural

STUDY DESIGN:
Intervention Model Description: All patients who accept participation in the study and meet all inclusion criteria will be randomly assigned at the time of anesthetic induction. The assignment to the group of epidural analgesia vs IV lidocaine will be 1: 1 randomly using permuted blocks generated by a computer operated by an external assistant to the investigation. The size of the blocks will be variable between 4, 6, and 8, and will be kept confidential to guarantee the concealment of the groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The masking process will be done as follows:
  Masking of the data collection and analysis staff: The investigative staff who performs the data collection and who evaluates the outcomes after the anesthetic act, will not have information about the intervention received by the patient. Those who participate in the data analysis phase will also be blind to the intervention.
  For practical and ethical point of view, it is not possible to mask the doctors who perform the intervention and neither the patients. A "SHAM" or simulated intervention is not possible given that this would require an unnecessary invasive procedure that would not be used, which would make it ethically questionable.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural Analgesia (Active Comparator): The placement of the thoracic epidural catheter will be located depending on surgical incision as follows:
  * Surgery of the upper abdomen: T7-T8.
  * Surgery of lower abdomen: T8-T9. The epidural catheter placement technique will be determined by the treating anesthesiologist. However, once the epidural space is located and the respective catheter is inserted, the correct location of the catheter should be tested with lidocaine at 2% CE 5 cc and a sensitivity test with temperature should be performed on the target dermatomes. A negative test for an adequate location of the catheter indicates that the procedure should be repeated until the epidural space is correctly located. Once this is achieved, the catheter will be left 4 cm away from the skin. The catheter will be fixed according to the institutional protocol.
  Interventions: Procedure: Epidural Analgesia
- Lidocaine Infussion (Experimental): Intravenous lidocaine
  Interventions: Drug: Lidocaine Infusion

INTERVENTIONS:
Procedure: Epidural Analgesia — The epidural infusion will be as follows:
  * Isobaric Bupivacaine 0.5% 40 cc
  * Morphine 4 mg (1 ampoule up to 10 cc and 4 cc of the mixture will be applied)
  * Saline solution 0.9% 156 cc.
  * Total Volume: 200 cc.
  This mixture will be prepared by a nurse outside the research group outside the operating room once indicated.
  The infusion will be scheduled at 7 cc / hour per continuous infusion set and will be connected to the epidural catheter after its placement.
  Arms: Epidural Analgesia
Drug: Lidocaine Infusion — 2% Lidocaine IV without epinephrine: 1 mg/kg/ hour for up to 24 hours, started immediately after anesthetic induction.
  Arms: Lidocaine Infussion

SUMMARY:
Major abdominal surgery continues is one of the most performed surgical procedures in the world, both electively and urgently. One of the main problems of this type of intervention is postoperative pain. it is shown that it increases health costs related to longer recovery times, longer hospital stay and related complications such as the increased risk of presenting chronic POP pain, which it has been estimated up to 20%, much higher if the surgery involves surgery in the gastrointestinal system.

The goal of analgesia in the postoperative setting is precisely to provide comfort to patients, minimize adverse effects and complications arising from the procedure.

The epidural analgesic technique (has been proposed as an analgesic management standard, since multiple studies have shown that it reduces opioid consumption, improves recovery and is a useful strategy for pain control. However, it is an invasive technique, with risk of complications such as hematomas and epidural abscesses, and it may be difficult to perform.

Currently it has been shown in multiple studies that the intravenous infusion of a local anesthetic, such as lidocaine, in this type of surgical scenarios can reduce the intensity of pain, opioid consumption, hospital stay and ileus with few adverse effects. In addition, these studies propose that, being a less invasive technique, it could be easier to implement and even be safer than the epidural technique.

The main hypothesis of this study is precisely that the infusion of lidocaine may be non-inferior to epidural analgesia in the analgesic management of patients undergoing major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years.
* Elective major open intra-abdominal surgery:

  * Cholecystectomy.
  * Total or subtotal gastrectomy.
  * Colectomy or Hemicolectomy.
  * Pancreatoduodenectomy.
  * Hepatectomy 1 or 2 segments.
  * Exploration and / or reconstruction of the bile duct.
  * Abdominal demolition.
  * Sigmoidectomy.
* Patient classified as ASA (American Association of Anesthesiology) 1, 2 or 3.

Exclusion Criteria:

* Pregnant woman
* Patient with contraindication for epidural analgesic techniques:

  1. Anticoagulated patient
  2. Active infection in the puncture site.
  3. Malformation in spinal cord.
  4. Sepsis without antibiotic treatment.
  5. Patient with contraindication for the use of intravenous lidocaine: Arrhythmias of any type not treated.
  6. Patient with known allergy to opioids and / or local anesthetics.
  7. Patient with chronic pain in previous management with strong opioids, gabapentinoids or epidural technique.
  8. Patient with liver failure or terminal renal failure.
  9. Patient who is scheduled for intubated admission to an intensive care unit after the procedure.
  10. Patient who refuses to participate in the study or who refuses to receive epidural analgesia.
  11. Patient who was technically impossible to place an epidural catheter in surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-09-05 (Actual); Study Completion 2022-09-05 (Actual)

PRIMARY OUTCOMES:
Posoperative Pain | 24 hours after surgery
  Numerical Rating Scale (NRS) for pain. The NRS for pain is a unidimensional measure of pain intensity in adults.The pain NRS is a single 11-point numeric scale. An 11-point numeric scale (NRS 11) with 0 representing one pain extreme (e.g., "no pain") and 10 representing the other pain extreme (e.g., "pain as bad as you can imagine" and "worst pain imaginable").

SECONDARY OUTCOMES:
Posoperative Pain | 2, 6, 12, 48 and 72 hours after surgery
  Numerical Rating Scale (NRS) for pain. The NRS for pain is a unidimensional measure of pain intensity in adults.The pain NRS is a single 11-point numeric scale. An 11-point numeric scale (NRS 11) with 0 representing one pain extreme (e.g., "no pain") and 10 representing the other pain extreme (e.g., "pain as bad as you can imagine" and "worst pain imaginable").
Posoperative opioid use | 24 hours after surgery
  mg of morphine
Hospital Stay | From date of randomization until the date day of discharge or date of death from any cause, whichever came first, assessed up to 100 months
  days
Perioperative Satisfaction | 24 hours
  Evaluation du Vecu de l'Anesthesie Generale (EVAN G scale). The EVAN questionnaire is composed of 6 dimensions (attention, privacy, information, pain, discomfort and waiting times), which in turn consist of 26 items. Each item is evaluated with in an ordinal scale. The minimum value is 1, meaning the worst value for the item and the maximum value is 5, meaning the better value for the item.
Toxicity by local anesthetics proportion | 24 hours after surgery
  Proportion of patients presenting signs of toxicity by local anesthetics.
  * Metal taste
  * Tinnitus
  * Hypotension (SBP less than 80 mmHg)
  * Tachycardia (FC greater than 130)
  * Bradycardia (FC less than 40)
  * Alterations of the mental state. It is positive for this outcome with 3 signs or if patient presents seizures or coma without a non-surgical or medical cause associated with the patient's clinical status.
Posoperative nausea and vomiting | 24 hours after surgey
  Proportion of patients with at least one episode of nausea or vomiting in the postoperative period.

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Casas, Dr, Principal Investigator — Univeridad de Antioquia's Professor
Locations (1):
- Antioquias Univervesity Health Institution, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shipton EA. The transition from acute to chronic post surgical pain. Anaesth Intensive Care. 2011 Sep;39(5):824-36. doi: 10.1177/0310057X1103900506. PMID 21970126
- [Result] Kranke P, Jokinen J, Pace NL, Schnabel A, Hollmann MW, Hahnenkamp K, Eberhart LH, Poepping DM, Weibel S. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery. Cochrane Database Syst Rev. 2015 Jul 16;(7):CD009642. doi: 10.1002/14651858.CD009642.pub2. PMID 26184397
- [Result] Couceiro TC, Valenca MM, Lima LC, de Menezes TC, Raposo MC. Prevalence and influence of gender, age, and type of surgery on postoperative pain. Rev Bras Anestesiol. 2009 May-Jun;59(3):314-20. doi: 10.1590/s0034-70942009000300006. English, Portuguese. PMID 19488544
- [Result] Singh PK, Saikia P, Lahakar M. Prevalence of acute post-operative pain in patients in adult age-group undergoing inpatient abdominal surgery and correlation of intensity of pain and satisfaction with analgesic management: A cross-sectional single institute-based study. Indian J Anaesth. 2016 Oct;60(10):737-743. doi: 10.4103/0019-5049.191686. PMID 27761037
- [Result] Bouman EA, Theunissen M, Bons SA, van Mook WN, Gramke HF, van Kleef M, Marcus MA. Reduced incidence of chronic postsurgical pain after epidural analgesia for abdominal surgery. Pain Pract. 2014 Feb;14(2):E76-84. doi: 10.1111/papr.12091. Epub 2013 Jun 12. PMID 23758753
- [Result] Li M, Li L, Xu Y, Wang X. Intravenous analgesics for pain management in post- operative patients : a comparative study of their efficacy and adverse effects. 2016;15(August):1799-806.
- [Result] Singh AP, Singh D, Singh Y, Jain G. Postoperative analgesic efficacy of epidural tramadol as adjutant to ropivacaine in adult upper abdominal surgeries. Anesth Essays Res. 2015 Sep-Dec;9(3):369-73. doi: 10.4103/0259-1162.161805. PMID 26712976
- [Result] Nworah U. From documentation to the problem: controlling postoperative pain. Nurs Forum. 2012 Apr-Jun;47(2):91-9. doi: 10.1111/j.1744-6198.2012.00262.x. PMID 22512766
- [Result] Sun Y, Li T, Wang N, Yun Y, Gan TJ. Perioperative systemic lidocaine for postoperative analgesia and recovery after abdominal surgery: a meta-analysis of randomized controlled trials. Dis Colon Rectum. 2012 Nov;55(11):1183-94. doi: 10.1097/DCR.0b013e318259bcd8. PMID 23044681
- [Result] Ventham NT, Kennedy ED, Brady RR, Paterson HM, Speake D, Foo I, Fearon KC. Efficacy of Intravenous Lidocaine for Postoperative Analgesia Following Laparoscopic Surgery: A Meta-Analysis. World J Surg. 2015 Sep;39(9):2220-34. doi: 10.1007/s00268-015-3105-6. PMID 26044546
- [Result] Kahokehr A, Sammour T, Soop M, Hill AG. Intraperitoneal local anaesthetic in abdominal surgery - a systematic review. ANZ J Surg. 2011 Apr;81(4):237-45. doi: 10.1111/j.1445-2197.2010.05573.x. Epub 2010 Nov 17. PMID 21418466
- [Result] Yu N, Long X, Lujan-Hernandez JR, Succar J, Xin X, Wang X. Transversus abdominis-plane block versus local anesthetic wound infiltration in lower abdominal surgery: a systematic review and meta-analysis of randomized controlled trials. BMC Anesthesiol. 2014 Dec 15;14:121. doi: 10.1186/1471-2253-14-121. eCollection 2014. PMID 25580086
- [Result] Ventham NT, Hughes M, O'Neill S, Johns N, Brady RR, Wigmore SJ. Systematic review and meta-analysis of continuous local anaesthetic wound infiltration versus epidural analgesia for postoperative pain following abdominal surgery. Br J Surg. 2013 Sep;100(10):1280-9. doi: 10.1002/bjs.9204. PMID 24244968
- [Result] Nimmo SM, Harrington LS. What is the role of epidural analgesia in abdominal surgery? Contin Educ Anaesthesia, Crit Care Pain. 2014;14(5):224-9.
- [Result] Nishimori M, Ballantyne JC, Low JH. Epidural pain relief versus systemic opioid-based pain relief for abdominal aortic surgery. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD005059. doi: 10.1002/14651858.CD005059.pub2. PMID 16856074
- [Result] Peters ML, Sommer M, de Rijke JM, Kessels F, Heineman E, Patijn J, Marcus MA, Vlaeyen JW, van Kleef M. Somatic and psychologic predictors of long-term unfavorable outcome after surgical intervention. Ann Surg. 2007 Mar;245(3):487-94. doi: 10.1097/01.sla.0000245495.79781.65. PMID 17435557
- [Result] Block BM, Liu SS, Rowlingson AJ, Cowan AR, Cowan JA Jr, Wu CL. Efficacy of postoperative epidural analgesia: a meta-analysis. JAMA. 2003 Nov 12;290(18):2455-63. doi: 10.1001/jama.290.18.2455. PMID 14612482
- [Result] Jorgensen H, Wetterslev J, Moiniche S, Dahl JB. Epidural local anaesthetics versus opioid-based analgesic regimens on postoperative gastrointestinal paralysis, PONV and pain after abdominal surgery. Cochrane Database Syst Rev. 2000;(4):CD001893. doi: 10.1002/14651858.CD001893. PMID 11034732
- [Result] Popping DM, Zahn PK, Van Aken HK, Dasch B, Boche R, Pogatzki-Zahn EM. Effectiveness and safety of postoperative pain management: a survey of 18 925 consecutive patients between 1998 and 2006 (2nd revision): a database analysis of prospectively raised data. Br J Anaesth. 2008 Dec;101(6):832-40. doi: 10.1093/bja/aen300. Epub 2008 Oct 22. PMID 18945716
- [Result] Terkawi AS, Tsang S, Kazemi A, Morton S, Luo R, Sanders DT, Regali LA, Columbano H, Kurtzeborn NY, Durieux ME. A Clinical Comparison of Intravenous and Epidural Local Anesthetic for Major Abdominal Surgery. Reg Anesth Pain Med. 2016 Jan-Feb;41(1):28-36. doi: 10.1097/AAP.0000000000000332. PMID 26650426
- [Result] Koppert W, Weigand M, Neumann F, Sittl R, Schuettler J, Schmelz M, Hering W. Perioperative intravenous lidocaine has preventive effects on postoperative pain and morphine consumption after major abdominal surgery. Anesth Analg. 2004 Apr;98(4):1050-1055. doi: 10.1213/01.ANE.0000104582.71710.EE. PMID 15041597
- [Result] Wongyingsinn M, Baldini G, Charlebois P, Liberman S, Stein B, Carli F. Intravenous lidocaine versus thoracic epidural analgesia: a randomized controlled trial in patients undergoing laparoscopic colorectal surgery using an enhanced recovery program. Reg Anesth Pain Med. 2011 May-Jun;36(3):241-8. doi: 10.1097/AAP.0b013e31820d4362. PMID 21519309
- [Result] Yardeni IZ, Beilin B, Mayburd E, Levinson Y, Bessler H. The effect of perioperative intravenous lidocaine on postoperative pain and immune function. Anesth Analg. 2009 Nov;109(5):1464-9. doi: 10.1213/ANE.0b013e3181bab1bd. PMID 19843784
- [Result] Staikou C, Avramidou A, Ayiomamitis GD, Vrakas S, Argyra E. Effects of intravenous versus epidural lidocaine infusion on pain intensity and bowel function after major large bowel surgery: a double-blind randomized controlled trial. J Gastrointest Surg. 2014 Dec;18(12):2155-62. doi: 10.1007/s11605-014-2659-1. Epub 2014 Sep 23. PMID 25245767
- [Result] Khan JS, Yousuf M, Victor JC, Sharma A, Siddiqui N. An estimation for an appropriate end time for an intraoperative intravenous lidocaine infusion in bowel surgery: a comparative meta-analysis. J Clin Anesth. 2016 Feb;28:95-104. doi: 10.1016/j.jclinane.2015.07.007. Epub 2015 Sep 3. PMID 26342631
- [Derived] Casas-Arroyave FD, Osorno-Upegui SC, Zamudio-Burbano MA. Therapeutic efficacy of intravenous lidocaine infusion compared with thoracic epidural analgesia in major abdominal surgery: a noninferiority randomised clinical trial. Br J Anaesth. 2023 Nov;131(5):947-954. doi: 10.1016/j.bja.2023.07.032. Epub 2023 Sep 26. PMID 37758623